CLINICAL TRIAL: NCT04831333
Title: Deep Learning-based System for Detection of AIDS-related Cytomegalovirus Retinitis in Ultra-Widefield Fundus Images
Brief Title: Deep Learning-based System and AIDS-related Cytomegalovirus Retinitis
Status: Completed | Type: Observational
Sponsor: Kuifang Du (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor-Investigator, Kuifang Du, Principal investigator, Beijing YouAn Hospital
Organization: Beijing YouAn Hospital (Other)
Other Study IDs: 20210331001
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cytomegalovirus Retinitis
Keywords: AIDS; HIV; Cytomegalovirus Retinitis; Deep learning; Ultra-wide-field imaging
MeSH Terms: conditions — Cytomegalovirus Retinitis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active CMVR: The UWF images of cytomegalovirus retinitis (CMVR) included various patterns: hemorrhagic necrotizing lesion, granular lesion, frosted branch angiitis, and optic neuropathy lesion. Active CMVR lesion was defined as obvious opacity (mild, moderate, severe, very severe)
- Inactive CMVR: Inactive CMVR lesion was defined as a lack of opacity or questionable/equivocal activity.
- Non-CMVR: The non-CMVR images included normal retina and other retinopathies such as HIV-related microvascular retinopathy, diabetic retinopathy, retinal detachment, vitreous hemorrhage.

INTERVENTIONS:
Other:

SUMMARY:
Ophthalmological screening for cytomegalovirus retinitis (CMVR) for HIV/AIDS patients is important. However, the manual screening with fundus imaging is laborious and subjective.

Deep learning (DL) system has been developed for the automated detection of various eye diseases with high accuracy and efficiency, including diabetic retinopathy, glaucoma, age-related macular degeneration (AMD), papilledema, lattice degeneration and retinal breaks, from ocular fundus photographs. UWF imaging is a relatively new imaging modality for DL system but has also shown extraordinary talents in automatic retinal analysis With the press for routine CMVR screening in AIDS patients and the great capacity of DL system, the use of deep learning (DL) system to AIDS-related CMVR with Ultra-Widefield (UWF) fundus images is promising.

The investigators previously developed a DL system to detect AIDS-related CMVR. For further evaluating the applicability of the DL system, a prospective dataset is needed.

ELIGIBILITY:
Inclusion Criteria:

The UWF images from HIV/AIDS patients.

Exclusion Criteria:

1. The UWF images would be excluded if all three human graders gave different diagnosis.
2. The UWF images with poor quality would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIDS patients undergoing OPTOS camera (OPTOS® Daytona) from Department of Ophthalmology, Beijing Youan Hospital, were prospectively collected as a prospective dataset.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluating the applicability of the DL system to identify AIDS-related CMVR | April 2021
  The investigators compared the performance between two trained (senior and junior) retinal ophthalmologists with the DL system. A senior retinal ophthalmologist and a junior retinal ophthalmologist were asked to independently screen the UWF images in the prospective dataset. Accuracy, sensitivity and specificity were used to evaluate the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Kui-Fang Du, Study Director — Beijing YouAn Hospital; Li Dong, Study Director — Beijing Tongren Hospital; Kai Zhang, Principal Investigator — Beijing Tongren Hospital; Chao Chen, Principal Investigator — Beijing YouAn Hospital; Lian-Yong Xie, Principal Investigator — Beijing YouAn Hospital; Wen-Jun Kong, Principal Investigator — Beijing YouAn Hospital; Hong-Wei Dong, Principal Investigator — Beijing YouAn Hospital; He-Yan Li, Principal Investigator — Beijing Tongren Hospital; Rui-Heng Zhang, Principal Investigator — Beijing Tongren Hospital; Wen-Da Zhou, Principal Investigator — Beijing Tongren Hospital; Hao-Tian Wu, Principal Investigator — Beijing Tongren Hospital; Wen-Bin Wei, Study Chair — Beijing Tongren Hospital
Locations (1):
- Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality, China